CLINICAL TRIAL: NCT02587962
Title: A Phase 1/2 Multicenter, Single-Arm, Open-Label, Dose-Escalation Study of Birinapant in Combination With Pembrolizumab (KEYTRUDA®) in Patients With Relapsed or Refractory Solid Tumors
Brief Title: Dose-escalation Study of Birinapant and Pembrolizumab in Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Based on a futility analysis, the data monitoring committee recommended to stop enrollment.
Sponsor: Medivir (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPT-201; MK3475 KEYNOTE KN163 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2015-10-21; First posted 2015-10-27 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2020-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — birinapant; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Birinapant in combination with pembrolizumab (Experimental): Birinapant in combination with pembrolizumab
  Interventions: Drug: Birinapant; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Birinapant — Birinapant intravenous (IV) on Days 1 and 8 of each 21-Day Cycle. The following escalating doses of birinapant to be studied: 5.6, 11, 17, and 22 mg/m2. In the expansion phase the assigned recommended phase two dose will be administered in all cohorts
Drug: Pembrolizumab — 200 mg pembrolizumab IV on Day 1 of each 21-Day Cycle
  Other Names: KEYTRUDA; lambrolizumab; MK-3475; SCH 9000475

SUMMARY:
An ascending dose study in patients with solid tumors to evaluate the safety, tolerability, pharmacodynamics and efficacy of birinapant when given in combination with pembrolizumab. A dose expansion phase of 4 cohorts will also be included.

DETAILED DESCRIPTION:
This study will be conducted in two phases. The Phase 1 portion of the study will employ a sequential group dose-escalation design to determine the dose-limiting toxicity (DLT) and recommended Phase 2 dose (RP2D) of birinapant administered in combination with 200 mg pembrolizumab, both administered as a 30-minute intravenous (IV) infusion. The following proposed doses of birinapant are to be evaluated: 5.6, 11, 17, and 22 mg/m2.

The Phase 2 portion, the dose expansion phase, will compromise 4 cohorts of 26-30 patients.

The 4 cohorts will include the following:

* Colorectal cancer
* Ovarian Cancer
* Cervical cancer
* Various solid tumors (30 patients, including 5 patients with each of the following 6 tumor types: Head and Neck Squamous Cell Carcinoma (HNSCC)-checkpoint-inhibitor naïve; and HNSCC checkpoint-inhibitor experienced; Gastroesophageal carcinoma; Mesothelioma; Small cell lung cancer (SCLC); Cholangiocarcinoma

A Simon's 2-stage design will be used for each of the cohorts in colorectal cancer, ovarian cancer and cervical cancer. A predefined interim analysis allowing stopping each of these cohorts for futility and safety will be conducted in the first stage to limit undue exposure before further inclusion into a given cohort. The design of the various solid tumors cohort will limit undue exposure in any of the selected tumor types by limiting the number of enrolled patient to five in each tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid malignancy that is metastatic or unresectable for which standard curative or palliative measures do not exist or are no longer effective (Dose Escalation phase only)
* Measurable disease according to response evaluation criteria in solid tumors (RECIST) v 1.1
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Normal organ and marrow function

Dose Expansion phase specific additional inclusion criteria:

* Patients with metastatic colorectal cancer with no available therapy options that are known to provide clinical benefit per institutional standard of care (colorectal cancer cohort only)
* Patients must have a histologically confirmed epithelial ovarian cancer, primary peritoneal cancer or fallopian tube solid tumor cancer that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care (ovarian cancer cohort only)
* Patients must have histologically or cytologically confirmed cervical squamous cell carcinoma that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care (cervical cancer cohort only)
* Patients must have histologically or cytologically confirmed head and neck squamous cell carcinoma that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care. (various solid tumors cohort: head and neck squamous cell carcinoma groups only).
* Patients must have received prior therapy with an anti-programmed death protein (PD-1) or anti-PD-ligand 1(L1) antibody, or previously participated in Merck MK 3475 clinical trials. Patients must have experienced documented, confirmed radiographic progression of disease by immune RECIST (iRECIST), or by RECIST v1.1 (various solid tumors cohort head and neck squamous cell carcinoma, Check point inhibitor experienced group only).
* Patients must have histologically or cytologically confirmed small cell lung carcinoma (SCLC) that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care (various solid tumors cohort, SCLC group only).
* Patients must have histologically or cytologically confirmed cholangiocarcinoma that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care (various solid tumors cohort, cholangiocarcinoma group only).
* Patients must have histologically or cytologically confirmed mesothelioma that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care (various solid tumors cohort, mesothelioma group only).
* Patients must have histologically or cytologically confirmed carcinoma of the esophagus including the gastroesophageal junction that is locally advanced or metastatic with no available therapy options that are known to provide clinical benefit per institutional standard of care (various solid tumors cohort, gastroesophageal carcinoma group only).

Exclusion Criteria:

Exclusion criteria apply to all phases and cohorts in the study unless otherwise stated

* Prior monoclonal antibody, within 4 weeks prior to first dose of study drug.
* Prior chemotherapy, targeted small molecule therapy or radiotherapy within 2 weeks prior to first dose of study drug.
* Patients who have received any other investigational agents within 4 weeks of first dose of study drug.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-ligand 2(L2), anti-cluster of differentiation 137 (anti-CD137), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody. (Not applicable for various solid tumors cohort, head and neck squamous cell carcinoma check-point inhibitor experienced group)
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to birinapant or pembrolizumab or their constituents.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, hypertension, unstable angina pectoris, cardiac arrhythmia, autoimmune disease or inflammatory diseases, or psychiatric illness/social situations that would limit compliance with study requirements.
* Evidence of active, non-infectious pneumonitis or a history of interstitial lung disease.
* Known history of Human Immunodeficiency Virus (HIV) (HIV1/2 antibodies), or Active Hepatitis B (HBsAg reactive). Patients with active Hepatitis C (HCV-RNA qualitative).
* Currently breast feeding, pregnant or planning to conceive or father Children from screening through 120 Days after last dose of study drug.
* Patients who have received anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) (Various solid tumor cohort, head and neck squamous cell carcinoma check point inhibitor experienced group only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Dept of Medicine-Hematology/Oncology, Santa Monica, California
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Thomas Jefferson University Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Mary Crowley Cancer Research, Dallas, Texas
  - MD Anderson Cancer Center, The University of Texas, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - 5.6 mg: Dose escalation (Phase 1): 5.6 mg birinapant + pembrolizumab
- Phase 1 - 11 mg: Dose escalation (Phase 1): 11 mg birinapant + pembrolizumab
- Phase 1 - 17 mg: Dose escalation (Phase 1): 17 mg birinapant + pembrolizumab
- Phase 1 - 22 mg: Dose escalation (Phase 1): 22 mg birinapant + pembrolizumab
- Phase 2 - 22 mg: Dose expansion (Phase 2): 22 mg birinapant + pembrolizumab
Period: Overall Study
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 - 22 mg
Started | 3 | 3 | 6 | 7 | 15
Completed (Completed study treatment phase) | 1 | 0 | 0 | 1 | 0
Not Completed | 2 | 3 | 6 | 6 | 15
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 4
Not completed — Radiological progression | 2 | 2 | 2 | 5 | 10
Not completed — Clinical progression | 0 | 1 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 - 22 mg | Total
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 15 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (16.09) | 71.3 (3.21) | 60.2 (6.15) | 59.1 (11.61) | 53.8 (10.43) | 60.08 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 4 | 10 | 23
  Male | 1 | 1 | 1 | 3 | 5 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 3 | 6 | 6 | 12 | 30
  Unknown | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6 | 7 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through blood pressure.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
mmHg
  Systolic blood pressure at baseline | 137.3 (18.6) | 143.3 (14.5) | 134.0 (22.1) | 118.6 (11.4)
  Systolic blood pressure at follow-up: number analyzed (Participants) | 1 | 2 | 3 | 1
  Systolic blood pressure at follow-up | 120.0 (NA) — Only 1 participant assessed at follow-up. | 107.0 (1.4) | 119.7 (30.2) | 120.0 (NA) — Only 1 participant assessed at follow-up.
  Diastolic blood pressure at baseline | 78.0 (2.0) | 77.0 (15.5) | 74.3 (9.3) | 66.6 (7.9)
  Diastolic blood pressure at follow-up: number analyzed (Participants) | 1 | 2 | 3 | 1
  Diastolic blood pressure at follow-up | 84.0 (NA) — Only 1 participant assessed at follow-up. | 66.0 (8.5) | 71.3 (11.4) | 75.0 (NA) — Only 1 participant assessed at follow-up.

2. Primary Outcome: Electrocardiogram: QT Interval (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through electrocardiogram.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
ms
  Electrocardiogram QT interval at baseline | 368.7 (30.6) | 388.3 (11.2) | 386.3 (32.9) | 365.9 (32.7)
  Electrocardiogram QT interval at follow-up: number analyzed (Participants) | 1 | 0 | 1 | 1
  Electrocardiogram QT interval at follow-up | 392.0 (NA) — Only 1 participant assessed at follow-up. |  | 380.0 (NA) — Only 1 participant assessed at follow-up. | 364.0 (NA) — Only 1 participant assessed at follow-up.

3. Primary Outcome: Amylase and Lipase (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through amylase and lipase.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
U/L
  Amylase at baseline | 33.7 (32.5) | 38.3 (9.0) | 64.3 (8.0) | 40.6 (27.4)
  Amylase at follow-up: number analyzed (Participants) | 1 | 2 | 2 | 1
  Amylase at follow-up | 27.0 (NA) — Only 1 participant assessed at follow-up. | 49.0 (41.0) | 56.5 (38.9) | 60.0 (NA) — Only 1 participant assessed at follow-up.
  Lipase at baseline | 17.0 (12.2) | 24.0 (21.0) | 32.2 (21.4) | 49.9 (63.3)
  Lipase at follow-up: number analyzed (Participants) | 1 | 2 | 2 | 7
  Lipase at follow-up | 12.0 (NA) — Only 1 participant assessed at follow-up. | 15.5 (10.6) | 16.0 (2.8) | 18.0 (NA) — Only 1 participant assessed at follow-up.

4. Primary Outcome: Thyroxine Free (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through thyroxine free.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
nmol/L
  Thyroxine free at baseline: number analyzed (Participants) | 2 | 2 | 6 | 7
  Thyroxine free at baseline | 16.8 (5.0) | 15.0 (3.0) | 15.0 (3.3) | 18.7 (1.6)
  Thyroxine free at last assessment: number analyzed (Participants) | 3 | 2 | 4 | 3
  Thyroxine free at last assessment | 25.2 (8.0) | 16.7 (5.4) | 16.9 (4.1) | 16.5 (3.6)

5. Primary Outcome: Thyrotropin (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through Thyrotropin.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
mU/L
  Thyrotropin at baseline: number analyzed (Participants) | 2 | 2 | 6 | 7
  Thyrotropin at baseline | 3.8 (3.2) | 2.4 (0.9) | 1.7 (0.8) | 1.4 (0.9)
  Thyrotropin at last assessment: number analyzed (Participants) | 3 | 3 | 4 | 3
  Thyrotropin at last assessment | 14.2 (18.7) | 7.7 (4.0) | 2.3 (1.3) | 2.6 (2.1)

6. Primary Outcome: Hemoglobin (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through hemoglobin.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
g/L
  Hemoglobin at baseline | 110.3 (20.2) | 107.3 (8.6) | 112.0 (11.8) | 102.0 (16.0)
  Hemoglobin at follow-up: number analyzed (Participants) | 1 | 2 | 2 | 1
  Hemoglobin at follow-up | 89.0 (NA) — Only 1 participant was assessed at follow-up | 107.0 (14.1) | 116.0 (19.8) | 99.0 (NA) — Only 1 participant was assessed at follow-up

7. Primary Outcome: Physical Exam (Safety and Tolerability in the Dose Escalation Phase)
Description: Evaluation of the safety and tolerability of birinapant when given in combination with pembrolizumab assessed through physical exam.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7
Participants
  Clinically significant physical exam abnormalities - baseline | 0 | 0 | 3 | 0
  Clinically significant physical exam abnormalities - last assessment: number analyzed (Participants) | 3 | 3 | 6 | 5
  Clinically significant physical exam abnormalities - last assessment | 0 | 1 | 3 | 0

8. Primary Outcome: Overall Response (Applicable for: Dose Escalation Phase and Dose Expansion Phase in Cohorts of Colorectal Cancer, Ovarian Cancer and Cervical Cancer)
Description: Evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. A responder was a patient who showed best overall response of complete response (CR, disappearance of all target lesions) or partial response (PR, ≥30% decrease in the sum of the longest diameter of target lesions), which was confirmed again at least 4 weeks after the initial assessment.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: For phase 2, only the colorectal cancer (CRC) cohort was analyzed for overall response rate. Patients were not recruited to the ovarian cancer or cervical cancer cohorts due to early termination of the study.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2 CRC - 22 mg: Dose expansion (Phase 2): 22 mg birinapant + pembrolizumab in colorectal cancer cohort.
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 15
Participants | 1 | 0 | 0 | 0 | 0

9. Secondary Outcome: Tumor Response Evaluated Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1:
Description: Analysis of progression-free survival (PFS); time to progression, where progressive disease (PD) corresponds to ≥20% increase in the sum of the longest diameter of target lesions.
Time Frame: Every 9 weeks; up to 2 yrs
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- Phase 2 CRC - 22 mg: Dose expansion (Phase 2): 22 mg birinapant + pembrolizumab
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 15
Weeks | 15.4 [11.3 to NA] — Due to low number of patients / lack of data, the upper inter-quartile could not be calculated. | 7.7 [4.0 to 9.6] | 8.6 [8.0 to 26.0] | 8.0 [4.1 to 8.9] | 9.0 [8.1 to 18.1]

10. Secondary Outcome: Blood Pressure (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of birinapant at the recommended phase 2 dose (RP2D) when given in combination with pembrolizumab assessed through blood pressure.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Phase 2 CRC - 22 mg: Dose expansion (Phase 2): 22 mg birinapant + pembrolizumab in colorectal cancer cohort (CRC)
Arm/Group | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 15
mmHg
  Systolic blood pressure at baseline | 130.9 (20.3)
  Systolic blood pressure at follow-up: number analyzed (Participants) | 9
  Systolic blood pressure at follow-up | 129.3 (16.6)
  Diastolic blood pressure at baseline | 80.0 (8.0)
  Diastolic blood pressure at follow-up: number analyzed (Participants) | 9
  Diastolic blood pressure at follow-up | 74.4 (12.2)

11. Secondary Outcome: Electrocardiogram: QT Interval (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of birinapant at the recommended phase 2 dose (RP2D) when given in combination with pembrolizumab assessed through electrocardiogram.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 15
ms
  Electrocardiogram QT interval at baseline | 383.5 (25.6)
  Electrocardiogram QT interval at follow-up: number analyzed (Participants) | 5
  Electrocardiogram QT interval at follow-up | 392.6 (38.7)

12. Secondary Outcome: Amylase and Lipase (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of birinapant at the recommended phase 2 dose (RP2D) when given in combination with pembrolizumab assessed through amylase and lipase.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 15
U/L
  Amylase at baseline | 68.9 (22.5)
  Amylase at follow-up: number analyzed (Participants) | 6
  Amylase at follow-up | 93.0 (35.4)
  Lipase at baseline | 44.3 (41.1)
  Lipase at follow-up: number analyzed (Participants) | 6
  Lipase at follow-up | 29.7 (16.6)

13. Secondary Outcome: Thyroxine Free (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of birinapant at the recommended phase 2 dose (RP2D) when given in combination with pembrolizumab assessed through thyroxine free.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 15
nmol/L
  Thyroxine free at baseline | 14.7 (3.1)
  Thyroxine free at last assessment: number analyzed (Participants) | 10
  Thyroxine free at last assessment | 16.4 (4.4)

14. Secondary Outcome: Thyrotropin (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of birinapant at the recommended phase 2 dose (RP2D) when given in combination with pembrolizumab assessed through thyrotropin.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 15
mU/L
  Thyrotropin at baseline | 2.3 (1.3)
  Thyrotropin at last assessment: number analyzed (Participants) | 12
  Thyrotropin at last assessment | 9.8 (23.5)

15. Secondary Outcome: Hemoglobin (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of birinapant at the recommended phase 2 dose (RP2D) when given in combination with pembrolizumab assessed through hemoglobin.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 15
g/L
  Hemoglobin at baseline | 126.4 (15.4)
  Hemoglobin at follow-up: number analyzed (Participants) | 13
  Hemoglobin at follow-up | 130.2 (13.2)

16. Secondary Outcome: Physical Exam (Safety and Tolerability in the Dose Expansion Phase - Colorectal Cancer Cohort)
Description: Evaluation of the safety and tolerability of the RP2D of birinapant when given in combination with pembrolizumab assessed through physical exam.
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: As the population of participants were very ill, assessments outside clinical praxis were sometimes not performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 - 22 mg
Number analyzed (Participants) | 15
Participants
  Clinically significant physical exam abnormalities - baseline | 0
  Clinically significant physical exam abnormalities - last assessment: number analyzed (Participants) | 14
  Clinically significant physical exam abnormalities - last assessment | 2

17. Other Pre Specified Outcome: Assess Tumor Activity
Description: To be evaluated according to immune response evaluation criteria in solid tumors (iRECIST)
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: Tumor activity according to iRECIST was not analyzed due to early termination of the study.
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

18. Other Pre Specified Outcome: Translational Biomarker Assessments Obtained From Blood
Description: Measured by inhibitor of apoptosis proteins (IAPs), cytokines, tumor infiltrating lymphocytes (TILs) cluster of differentiation (CD)3, CD4, CD8, and CD19 as well as absolute neutrophil and lymphocyte counts
Time Frame: Day 1 through Day 8
Population: Biomarkers in blood were not analyzed due to early termination of the study.
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Other Pre Specified Outcome: Translational Biomarker Assessments of Tumor Biopsy Samples
Description: Measured by: Programmed death ligand 1 (PD-1L), programmed cell death protein 1 receptor (PD-1) and related proteins, genome analysis, IAP gene copy number and TILs cluster of differentiation (CD)3, CD4, CD8 and CD19
Time Frame: Baseline and up to 2 yrs (follow-up)
Population: Biomarkers in tumor biopsy samples were not analyzed due to early termination of the study.
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Other Pre Specified Outcome: Pharmacokinetics of Birinapant in Plasma
Description: The plasma concentrations of birinapant was to be measured and summarized descriptively
Time Frame: Day 1 through Day 8
Population: Birinapant pharmacokinetics was not analyzed due to early termination of the study.
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Phase 1 - 5.6 mg | Phase 1 - 11 mg | Phase 1 - 17 mg | Phase 1 - 22 mg | Phase 2 CRC - 22 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 0/7 | 1/15
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 4/6 | 3/7 | 5/15
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 7/7 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - 5.6 mg (N=3) | Phase 1 - 11 mg (N=3) | Phase 1 - 17 mg (N=6) | Phase 1 - 22 mg (N=7) | Phase 2 CRC - 22 mg (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — The event leading to death (the underlying cause) was unknown and therefore reported by the Investigator as preferred term 'Death'
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Smal intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 - 5.6 mg (N=3) | Phase 1 - 11 mg (N=3) | Phase 1 - 17 mg (N=6) | Phase 1 - 22 mg (N=7) | Phase 2 CRC - 22 mg (N=15)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 5 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 2 (5) | 2 (4) | 4 (7)
Weight increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Gastric hypomotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic failure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (4) | 3 (8) | 3 (4)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (8)
Foreign body sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyposmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Bloody discharge (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (5)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinaemia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (11)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroxine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The dose escalation (Phase 1) part was analyzed per the protocol. Based on data from the interim analysis of the colorectal cancer cohort (dose expansion [Phase 2] part), the study was closed early due to futility on recommendation by the data monitoring committee (DMC).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must submit any proposed publication or presentation to the Sponsor, along with information about the scientific journal or presentation forum, at least 30 days before submission of the publication or presentation (2 weeks for abstracts). The Investigator will comply with Sponsor requests to delete confidential information (other than the study results) and to withhold publication or presentation for an additional 60 days in order to obtain patent protection if necessary.

DOCUMENTS (2):
  • Study Protocol (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT02587962/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT02587962/SAP_001.pdf